CLINICAL TRIAL: NCT01160822
Title: A Randomized, Double Blind, Placebo and Naproxen Controlled, Multi-center, Study to Determine the Safety, Tolerability, Pharmacokinetics and Effect on Pain of a Single Intra-articular Administration of Canakinumab in Patients With Osteoarthritis in the Knee
Brief Title: To Determine the Safety, Tolerability, Pharmacokinetics and Effect on Pain of a Single Intra-articular Administration of Canakinumab in Patients With Osteoarthritis in the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CACZ885C2201; 2009-015017-48 (EudraCT Number)
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Results first posted 2012-08-30 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-09

CONDITIONS: Osteoarthritis
Keywords: Osteo arthritis; pain control; intra- articular injections; Knee OA
MeSH Terms: conditions — Osteoarthritis; Agnosia | interventions — canakinumab; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (5):
- Part A: Canakinumab (Experimental): In this ascending dose part, participants received a single intra-articular injection of canakinumab. The beginning dose was 150 mg, escalating to the 300 mg dose and then to 600 mg.
  Interventions: Biological: Canakinumab
- Part A: Placebo (Placebo Comparator): Participants received a single intra-articular injection of canakinumab-matching placebo.
  Interventions: Drug: Placebo to canakinumab
- Part B: Canakinumab (Experimental): Participants received a single intra-articular injection of canakinumab on Day 1 and naproxen matching placebo tablets orally twice daily for 12 weeks.
  Interventions: Biological: Canakinumab; Drug: Placebo to Naproxen
- Part B: Placebo (Placebo Comparator): Participants received a single intra-articular injection of canakinumab matching placebo on Day 1 and naproxen matching placebo tablets orally twice daily for 12 weeks.
  Interventions: Drug: Placebo to canakinumab; Drug: Placebo to Naproxen
- Part B: Naproxen (Active Comparator): Participants received a single intra-articular injection of canakinumab matching placebo on Day 1 and naproxen 500mg tablets orally twice daily for 12 weeks.
  Interventions: Drug: Placebo to canakinumab; Drug: Naproxen

INTERVENTIONS:
Biological: Canakinumab — Intra-articular injection
  Other Names: ACZ885
  Arms: Part A: Canakinumab; Part B: Canakinumab
Drug: Placebo to canakinumab — Intra-articular injection
  Arms: Part A: Placebo; Part B: Naproxen; Part B: Placebo
Drug: Naproxen — Tablets for oral administration
  Arms: Part B: Naproxen
Drug: Placebo to Naproxen — Tablets for oral administration
  Arms: Part B: Canakinumab; Part B: Placebo

SUMMARY:
The purpose of this study was to determine whether, in patients with mild to moderate knee osteoarthritis, canakinumab is safe and tolerable when injected intra-articularly.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel group, placebo controlled 18 weeks study, consisting of two parts:

1. Part A: an ascending single dose part in which the safety and tolerability of up to 4 different canakinumab doses are studied (starting dose 150 mg, maximum dose 600 mg).
2. Part B: a double-dummy, active-controlled, parallel design part in which the pain reduction of the canakinumab dose selected from part A is studied in comparison to Placebo and Naproxen.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Male and female patients aged 40 - 80 years (inclusive).
3. Diagnosis of knee osteoarthritis
4. Radiographic evidence of tibiofemoral compartment osteoarthritis
5. Pain in the knee during the last 24 hours.The patients should also have had pain in the affected knee on most days over the last month.
6. Patients who are willing to discontinue all non-steroidal anti-inflammatory drugs (NSAIDs) or other analgesic medication taken for any condition, including their knee pain,
7. Patients who are on stable dose of opioids for at least 1 month before screening can continue to take their opioid at this stable dose throughout the study.
8. Patients must also be willing to abstain from any intra-articular or peri-articular injections to the knee or surgery during the treatment period
9. Patients who, if they are currently taking aspirin (325 mg/day or less; as anti-coagulants), are willing to remain on a stable dose one month prior to screening and throughout the study

Exclusion Criteria:

1. Subjects with known hypersensitivity to any biological or investigational drugs.
2. Patients with contraindications to knee injections
3. Patients with joint effusion
4. Patients should not have rheumatoid arthritis or any connective tissue like disease
5. Secondary osteoarthritis with history and/or any evidence of the following diseases: septic arthritis, inflammatory joint disease, gout, Paget's disease of the bone, articular fracture, major dysplasias or congenital abnormality, ochronosis, acromegaly, hemochromatosis, Wilson's disease, primary osteochondromatosis, juvenile chronic arthritis with continued activity in adulthood, heritable disorders (e.g. hypermobility). Patients with secondary osteoarthritis following menisectomy or injuries of a collateral or cruciate ligament are not excluded.
6. Presence or history of underlying metabolic, endocrine, hematologic, pulmonary, cardiac, blood, renal, hepatic, infectious, psychiatric or gastrointestinal conditions
7. Evidence of tuberculosis (TB)
8. One of the risk factors for TB such as:

   1. Substance abuse (e.g. injection or non-injection)
   2. Health-care workers with unprotected exposure to patients who are at high risk of TB
   3. Patients with TB disease before the identification and correct airborne precautions of the patient
   4. close contact (i.e. share the same air space in a household or other enclosed environment for a prolonged period (days or weeks, not minutes or hours)) with a person with active pulmonary TB disease.
9. Significant medical problems, including but not limited to the following: uncontrolled hypertension,congestive heart failure, uncontrolled diabetes type I and II
10. Subjects with evidence of hepatic or blood coagulation disorders (i.e. hemophilia, etc), anemia, idiopathic thrombocytopenic purpura, or gastrointestinal disorder: severe hepatic disease, history of alcohol and drug abuse; disease of gall bladder and pancreas; active peptic ulceration, gastrointestinal bleeding or history of severe gastro-esophageal reflux disease or severe hiatus hernia; inflammatory bowel disease.
11. Use of any therapeutic protein drug (e.g. anti-tumor necrosis factor alpha (TNFα) antibody)
12. Presence of severe renal function impairment. History of renal trauma, glomerulonephritis, patients with one kidney, or renal failure requiring regular dialysis treatment.
13. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive pregnancy test (serum or urine).
14. Subjects with known contra-indications to naproxen (e.g. heart or circulation problems, history of ulcer disease etc.), analgesics, antipyretics, or NSAIDs.
15. Disease of the spine or other lower extremity joints which may interfere with the assessment of the target joint.
16. Surgery on the knee within the last year. Observational arthroscopy, arthroscopic surgery or lavage of the knee within the last 6 months.
17. Use of assistive devices other than a cane (walking stick) or knee brace.
18. Subjects who have experienced, any time in the past, asthma, acute rhinitis, nasal polyps, angioneurotic edema, urticaria or other allergic-type reaction after taking acetylsalicylic acid (ASA)/ aspirin or NSAIDs.
19. Any history of prior peptic ulcer disease or prior NSAID gastrointestinal complications for the past 5 years.

Other protocol defined inclusion/exclusion criteria may apply.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2010-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- United States (8):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Arizona Arthritis & Rheumatology Research, PLLC, Mesa, Arizona
  - San Diego Arthritis & Osteoporosis Medical Clinic, San Diego, California
  - Westlake Medical Research, Westlake Village, California
  - Rush-Presbyterian St. Lukes Medical Center, Chicago, Illinois
  - Cotton O'Neil Clinical Research Institute, Topeka, Kansas
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Volunteer Research Group, Knoxville, Tennessee
- Finland (2):
  - Novartis Investigative site, Helsinki
  - Novartis Investigative site, Kuopio
- Novartis Investigative site, Créteil, France
- Germany (2):
  - Novartis Investigative site, Berlin
  - Novartis Investigative site, Erlangen

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Canakinumab 150 mg: Participants received a single intra-articular injection of 150 mg canakinumab.
- Part A: Canakinumab 300 mg: Participants received a single intra-articular injection of 300 mg canakinumab.
- Part A: Canakinumab 600 mg: Participants received a single intra-articular injection of 600 mg canakinumab.
- Part B: Canakinumab: Participants received a single intra-articular injection of 600 mg canakinumab on Day 1 and naproxen matching placebo tablets orally twice daily for 12 weeks.
Period: Overall Study
Arm/Group | Part A: Canakinumab 150 mg | Part A: Canakinumab 300 mg | Part A: Canakinumab 600 mg | Part A: Placebo | Part B: Canakinumab | Part B: Placebo | Part B: Naproxen
Started | 6 | 7 | 6 | 5 | 45 | 47 | 53
Completed | 6 | 7 | 6 | 5 | 36 | 40 | 44
Not Completed | 0 | 0 | 0 | 0 | 9 | 7 | 9
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 2 | 5
Not completed — Unsatisfactory therapeutic effect | 0 | 0 | 0 | 0 | 4 | 5 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Administrative problems | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol deviation | 0 | 0 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Canakinumab 150 mg | Part A: Canakinumab 300 mg | Part A: Canakinumab 600 mg | Part A: Placebo | Part B: Canakinumab | Part B: Placebo | Part B: Naproxen | Total
Number analyzed (Participants) | 6 | 7 | 6 | 5 | 45 | 47 | 53 | 169
Age Continuous [Mean (Standard Deviation); unit: years] | 58.3 (12.79) | 61.0 (9.63) | 64.2 (10.68) | 57.8 (7.76) | NA (NA) — Age demographic data for Study Part A. | NA (NA) — Age demographic data for Study Part A. | NA (NA) — Age demographic data for Study Part A. | 60.5 (10.07)
Age, Customized [Mean (Standard Deviation); unit: years] | NA (NA) — Age demographic data for Study Part B. | NA (NA) — Age demographic data for Study Part B. | NA (NA) — Age demographic data for Study Part B. | NA (NA) — Age demographic data for Study Part B. | 61.4 (8.96) | 60.3 (9.71) | 62.2 (8.10) | 61.3 (8.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 2 | 2 | 31 | 31 | 34 | 107
  Male | 3 | 3 | 4 | 3 | 14 | 16 | 19 | 62

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Intolerance Events
Description: An intolerance event is defined as an acute inflammatory reaction, characterized by a 30 mm increase in pain (on a 100 mm visual analog scale (VAS) and associated with a new or worsened synovial fluid effusion within 3 days following the intra-articular (i.a.) injection. If baseline VAS pain score is ≥ 70 mm, an intolerance event is defined as an increase in pain by 20 mm on a 100 mm VAS associated with new or worsened synovial fluid effusion within 3 days following the i.a. injection. If baseline VAS pain score is ≥ 80 mm, an intolerance event is defined as an increase in pain by 10 mm on a 100 mm VAS associated with new or worsened synovial fluid effusion within 3 days following the i.a. injection. If baseline pain score is ≥ 90 mm, an intolerance event is defined as the patients experiencing an unspecified increase in pain on a 100 mm VAS associated with new or worsened synovial fluid effusion within 3 days following the i.a. injection.
Time Frame: Baseline to Day 3
Population: Safety analysis set.
Measure: Number; unit: participants
Arm/Group | Part A: Canakinumab 150 mg | Part A: Canakinumab 300 mg | Part A: Canakinumab 600 mg | Part A: Placebo
Number analyzed (Participants) | 6 | 7 | 6 | 5
participants | 0 | 0 | 0 | 0

2. Primary Outcome: Part B: Change From Baseline to Day 4 in Pain Using 100 mm Visual Analog Scale (VAS)
Description: After walking for 20 meters, participants were asked to assess the pain in their affected knee on a 100 mm linear visual analog scale ranging from no pain (0 mm) to unbearable pain (100 mm). A negative change from Baseline score indicates improvement.
  Results are from a Bayesian analysis of covariance (ANCOVA) model, fitting baseline pain VAS score as a covariate, time by treatment as fixed effects, region and subject as random effects.
Time Frame: Baseline and Day 4
Population: Pharmacodynamic (PD) analysis set - Patients with any available PD data and no major protocol deviations with impact on PD data, and where data were available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part B: Canakinumab | Part B: Placebo | Part B: Naproxen
Number analyzed (Participants) | 42 | 44 | 49
units on a scale | -26.7 (4.05) | -26.5 (3.97) | -27.6 (3.82)

3. Primary Outcome: Part B: Change From Baseline to Week 4 in Western Ontario and McMaster Osteoarthritis Index (WOMAC) Pain Subscale
Description: The Western Ontario and McMaster osteoarthritis Index (WOMAC) pain subscale asks patients to rate pain in the index knee joint in the last 48 hours doing different activities on a scale from none (0) to extreme pain (4). The answers are summed and the total pain subscale score ranges from 0 to 20, where higher scores indicate more pain. A negative change from Baseline score indicates improvement.
  Results are from a Bayesian ANCOVA model, fitting baseline WOMAC pain score as a covariate, time by treatment as fixed effects, region and patient as random effects.
Time Frame: Baseline and Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part B: Canakinumab | Part B: Placebo | Part B: Naproxen
Number analyzed (Participants) | 42 | 44 | 48
units on a scale | -3.5 (0.71) | -4.0 (0.68) | -4.5 (0.65)

4. Secondary Outcome: Part B: Change From Baseline in Pain Using 100 mm Visual Analog Scale (VAS)
Description: After walking for 20 meters, participants were asked to assess the pain in their affected knee on a 100 mm linear visual analog scale ranging from no pain (0 mm) to unbearable pain (100 mm).
  Results are from a Bayesian ANCOVA model, fitting baseline pain VAS score as a covariate, time by treatment as fixed effects, region and patient as random effects.
Time Frame: Baseline and Weeks 4, 8 and 12
Population: Pharmacodynamic (PD) analysis set - Patients with any available PD data and no major protocol deviations with impact on PD data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part B: Canakinumab | Part B: Placebo | Part B: Naproxen
Number analyzed (Participants) | 43 | 44 | 49
units on a scale
  Week 4 | -25.6 (4.03) | -31.1 (4.03) | -36.1 (3.84)
  Week 8 | -26.2 (4.12) | -30.9 (4.06) | -33.0 (3.89)
  Week 12 | -25.1 (4.14) | -32.1 (4.06) | -27.8 (3.94)

5. Secondary Outcome: Part B: Percentage of Responders in the Pain 100 mm Visual Analog Scale (VAS)
Description: A responder is defined as a participant with a 50% or greater reduction from baseline on the VAS scale for pain assessment. After walking for 20 meters, participants were asked to assess the pain in their affected knee on a 100 mm linear visual analog scale ranging from no pain (0 mm) to unbearable pain (100 mm).
Time Frame: Baseline, Day 4, Weeks 1, 2, 4, 8 and 12
Population: Pharmacodynamic (PD) analysis set - Patients with any available PD data and no major protocol deviations with impact on PD data. N is the number of participants with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Canakinumab | Part B: Placebo | Part B: Naproxen
Number analyzed (Participants) | 43 | 44 | 49
percentage of participants
  Day 4 [N=42, 44, 48] | 50.0 | 43.2 | 47.9
  Week 1 [N=42, 44, 48] | 40.5 | 45.5 | 56.3
  Week 2 [N=41, 44, 48] | 46.3 | 43.2 | 62.5
  Week 4 [N=39, 40, 46] | 51.3 | 55.0 | 71.7
  Week 8 [N=36, 38, 43] | 52.8 | 50.0 | 55.8
  Week 12 [N=35, 37, 41] | 48.6 | 51.4 | 53.7

6. Secondary Outcome: Part B: Change From Baseline in WOMAC Pain, Stiffness and Physical Function Subscales
Description: The WOMAC consists of 3 subscales:
  The Pain subscale asks patients to rate pain in the index knee joint in the last 48 hours during walking, using stairs, in bed, sitting or lying, and standing on a scale from none (0) to extreme pain (4). The answers are summed and the total pain subscale score ranges from 0-20.
  The Stiffness subscale assesses stiffness in the index knee joint during the last 48 hours doing different activities on a scale from none (0) to extreme stiffness (4). The total stiffness subscale score ranges from 0-8.
  The Physical Function subscale assesses difficulty performing daily physical activities during the last 48 hours on a scale from none (0) to extreme difficulty (4). The total physical function subscale score ranges from 0-68.
  Higher scores indicate more pain/stiffness/difficulty. Results are from a Bayesian ANCOVA model, with baseline WOMAC score as a covariate, time by treatment as fixed effects, region and patient as random effects.
Time Frame: Baseline and Weeks 4, 8 and 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part B: Canakinumab | Part B: Placebo | Part B: Naproxen
Number analyzed (Participants) | 43 | 44 | 49
units on a scale
  Pain at Week 8 | -3.7 (0.72) | -4.2 (0.69) | -4.6 (0.66)
  Pain at Week 12 | -3.2 (0.72) | -4.5 (0.69) | -4.0 (0.66)
  Stiffness at Week 4 | -1.3 (0.36) | -1.5 (0.36) | -1.9 (0.34)
  Stiffness at Week 8 | -1.3 (0.37) | -1.5 (0.36) | -2.0 (0.35)
  Stiffness at Week 12 | -1.1 (0.37) | -1.7 (0.37) | -1.4 (0.35)
  Function at Week 4 [N=38, 39, 43] | -14.1 (1.93) | -15.9 (1.93) | -16.2 (1.76)
  Function at Week 8 [N=35, 36, 41] | -13.7 (1.97) | -14.9 (1.94) | -16.1 (1.77)
  Function at Week 12 [N= 33, 36, 39] | -13.4 (2.01) | -16.5 (1.96) | -14.4 (1.80)

7. Secondary Outcome: Part B: Proportion of Participants Who Used Rescue Analgesic During Study
Description: Participants were permitted to take oral rescue medication (Acetaminophen ≤ 4 gram/day) up until 24 hours of a scheduled assessment visit during the 12-week treatment period. The estimates shown are the Kaplan-Meier estimates of the proportion of participants that took rescue medication.
Time Frame: Day 4, Weeks 1, 2, 4, 8 and 12
Population: Safety analysis set (all participants as assigned that received at least one dose of study drug).
Measure: Number; unit: proportion of participants
Arm/Group | Part B: Canakinumab | Part B: Placebo | Part B: Naproxen
Number analyzed (Participants) | 45 | 47 | 53
proportion of participants
  Day 4 | 0.27 | 0.30 | 0.19
  Week 1 | 0.45 | 0.47 | 0.23
  Week 2 | 0.52 | 0.57 | 0.33
  Week 4 | 0.55 | 0.60 | 0.43
  Week 8 | 0.57 | 0.69 | 0.59
  Week 12 | 0.62 | 0.75 | 0.70

8. Secondary Outcome: Patient's Global Assessment of Response to Treatment on Day 4
Description: Participants made a global assessment of their response to treatment using a 5-point Likert scale: Excellent, Good, Acceptable, Poor, Very Poor.
Time Frame: Day 4
Population: Pharmacodynamic analysis set, where data were available.
Measure: Number; unit: participants
Arm/Group | Part B: Canakinumab | Part B: Placebo | Part B: Naproxen
Number analyzed (Participants) | 42 | 44 | 48
participants
  Excellent | 6 | 8 | 4
  Good | 14 | 16 | 20
  Acceptable | 11 | 13 | 16
  Poor | 5 | 5 | 6
  Very poor | 6 | 2 | 2

9. Secondary Outcome: Patient's Global Assessment of Response to Treatment at Week 2
Description: as for outcome 8
Time Frame: Week 2
Population: Pharmacodynamic analysis set, where data were available.
Measure: Number; unit: participants
Arm/Group | Part B: Canakinumab | Part B: Placebo | Part B: Naproxen
Number analyzed (Participants) | 41 | 43 | 48
participants
  Excellent | 5 | 6 | 11
  Good | 12 | 16 | 19
  Acceptable | 13 | 14 | 12
  Poor | 9 | 5 | 5
  Very poor | 2 | 2 | 1

10. Secondary Outcome: Patient's Global Assessment of Response to Treatment at Week 4
Description: as for outcome 8
Time Frame: Week 4
Population: Pharmacodynamic analysis set, where data were available.
Measure: Number; unit: participants
Arm/Group | Part B: Canakinumab | Part B: Placebo | Part B: Naproxen
Number analyzed (Participants) | 39 | 40 | 46
participants
  Excellent | 5 | 6 | 9
  Good | 15 | 16 | 18
  Acceptable | 10 | 10 | 13
  Poor | 8 | 6 | 4
  Very poor | 1 | 2 | 2

11. Secondary Outcome: Patient's Global Assessment of Response to Treatment at Week 8
Description: as for outcome 8
Time Frame: Week 8
Population: Pharmacodynamic analysis set, where data were available.
Measure: Number; unit: participants
Arm/Group | Part B: Canakinumab | Part B: Placebo | Part B: Naproxen
Number analyzed (Participants) | 36 | 38 | 43
participants
  Excellent | 5 | 5 | 10
  Good | 9 | 19 | 18
  Acceptable | 11 | 8 | 9
  Poor | 9 | 5 | 5
  Very poor | 2 | 1 | 1

12. Secondary Outcome: Patient's Global Assessment of Response to Treatment at Week 12
Description: as for outcome 8
Time Frame: Week 12
Population: Pharmacodynamic analysis set, where data were available.
Measure: Number; unit: participants
Arm/Group | Part B: Canakinumab | Part B: Placebo | Part B: Naproxen
Number analyzed (Participants) | 35 | 37 | 41
participants
  Excellent | 4 | 8 | 7
  Good | 12 | 13 | 15
  Acceptable | 7 | 14 | 13
  Poor | 11 | 2 | 5
  Very poor | 1 | 0 | 1

13. Secondary Outcome: Part B: Physician's Global Assessment of Response to Treatment at Day 4
Description: The study physician made a global assessment of response to treatment using a 5-point Likert scale: Excellent, Good, Acceptable, Poor, Very Poor.
Time Frame: Day 4
Population: Pharmacodynamic analysis set, where data were available.
Measure: Number; unit: participants
Arm/Group | Part B: Canakinumab | Part B: Placebo | Part B: Naproxen
Number analyzed (Participants) | 42 | 44 | 48
participants
  Excellent | 8 | 7 | 6
  Good | 11 | 18 | 21
  Acceptable | 16 | 14 | 13
  Poor | 4 | 3 | 7
  Very poor | 3 | 2 | 1

14. Secondary Outcome: Part B: Physician's Global Assessment of Response to Treatment at Week 2
Description: as for outcome 13
Time Frame: Week 2
Population: Pharmacodynamic analysis set, where data were available.
Measure: Number; unit: participants
Arm/Group | Part B: Canakinumab | Part B: Placebo | Part B: Naproxen
Number analyzed (Participants) | 40 | 44 | 48
participants
  Excellent | 7 | 5 | 15
  Good | 15 | 20 | 20
  Acceptable | 10 | 13 | 9
  Poor | 6 | 4 | 4
  Very poor | 2 | 2 | 0

15. Secondary Outcome: Part B: Physician's Global Assessment of Response to Treatment at Week 4
Description: as for outcome 13
Time Frame: Week 4
Population: Pharmacodynamic analysis set, where data were available.
Measure: Number; unit: participants
Arm/Group | Part B: Canakinumab | Part B: Placebo | Part B: Naproxen
Number analyzed (Participants) | 39 | 40 | 46
participants
  Excellent | 4 | 5 | 9
  Good | 15 | 20 | 21
  Acceptable | 14 | 11 | 12
  Poor | 5 | 3 | 4
  Very poor | 1 | 1 | 0

16. Secondary Outcome: Part B: Physician's Global Assessment of Response to Treatment at Week 8
Description: as for outcome 13
Time Frame: Week 8
Population: Pharmacodynamic analysis set, where data were available.
Measure: Number; unit: participants
Arm/Group | Part B: Canakinumab | Part B: Placebo | Part B: Naproxen
Number analyzed (Participants) | 36 | 38 | 43
participants
  Excellent | 5 | 3 | 9
  Good | 13 | 22 | 16
  Acceptable | 10 | 11 | 13
  Poor | 7 | 2 | 5
  Very poor | 1 | 0 | 0

17. Secondary Outcome: Part B: Physician's Global Assessment of Response to Treatment at Week 12
Description: as for outcome 13
Time Frame: Week 12
Population: Pharmacodynamic analysis set, where data were available.
Measure: Number; unit: participants
Arm/Group | Part B: Canakinumab | Part B: Placebo | Part B: Naproxen
Number analyzed (Participants) | 35 | 37 | 41
participants
  Excellent | 5 | 7 | 10
  Good | 13 | 16 | 15
  Acceptable | 6 | 12 | 8
  Poor | 9 | 2 | 7
  Very poor | 2 | 0 | 1

18. Secondary Outcome: Maximum Observed Plasma Concentration of Canakinumab (Cmax)
Time Frame: Day 1, pre-dose and 1, 3, 6 and 8 hours post-dose (Part A only), Day 2, 4, 8, 15, 29, 57, 85 and 126.
Population: Pharmacokinetic analysis set where data were available.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Part A: Canakinumab 150 mg | Part A: Canakinumab 300 mg | Part A: Canakinumab 600 mg | Part B: Canakinumab
Number analyzed (Participants) | 6 | 6 | 6 | 39
µg/mL | 23.0 (8.54) | 34.8 (11.3) | 65.5 (14.5) | 77.8 (22.8)

19. Secondary Outcome: Time to Reach the Maximum Observed Plasma Concentration of Canakinumab (Tmax)
Time Frame: Day 1, pre-dose and 1, 3, 6 and 8 hours post-dose (Part A only), Day 2, 4, 8, 15, 29, 57, 85 and 126.
Population: Pharmacokinetic analysis set where data were available.
Measure: Median (Full Range); unit: hours
Arm/Group | Part A: Canakinumab 150 mg | Part A: Canakinumab 300 mg | Part A: Canakinumab 600 mg | Part B: Canakinumab
Number analyzed (Participants) | 6 | 6 | 6 | 39
hours | 96.2 [74.6 to 164] | 86.7 [71.8 to 174] | 144 [71.5 to 197] | 95.9 [46.3 to 335]

20. Secondary Outcome: Area Under the Concentration Time Curve up to the Last Measurable Concentration (AUClast)
Time Frame: Day 1, pre-dose and 1, 3, 6 and 8 hours post-dose (Part A only), Day 2, 4, 8, 15, 29, 57, 85 and 126.
Population: Pharmacokinetic analysis set where data were available.
Measure: Mean (Standard Deviation); unit: µg*day/mL
Arm/Group | Part A: Canakinumab 150 mg | Part A: Canakinumab 300 mg | Part A: Canakinumab 600 mg | Part B: Canakinumab
Number analyzed (Participants) | 6 | 6 | 6 | 35
µg*day/mL | 16900 (4430) | 30700 (8380) | 56100 (23900) | 71900 (23800)

21. Secondary Outcome: Area Under the Concentration Time Curve From Time Zero to Infinity AUC(0-inf)
Time Frame: Day 1, pre-dose and 1, 3, 6 and 8 hours post-dose (Part A only), Day 2, 4, 8, 15, 29, 57, 85 and 126.
Population: Pharmacokinetic analysis set where data were available.
Measure: Mean (Standard Deviation); unit: µg*day/mL
Arm/Group | Part A: Canakinumab 150 mg | Part A: Canakinumab 300 mg | Part A: Canakinumab 600 mg | Part B: Canakinumab
Number analyzed (Participants) | 5 | 6 | 5 | 33
µg*day/mL | 16900 (4780) | 32400 (8010) | 49300 (16100) | 78300 (28000)

22. Secondary Outcome: Terminal Phase Half-life (t1/2) of Canakinumab
Description: The time it takes for the concentration level of canakinumab to fall to 50% of the original value.
Time Frame: Day 1, pre-dose and 1, 3, 6 and 8 hours post-dose (Part A only), Day 2, 4, 8, 15, 29, 57, 85 and 126.
Population: Pharmacokinetic analysis set where data were available.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part A: Canakinumab 150 mg | Part A: Canakinumab 300 mg | Part A: Canakinumab 600 mg | Part B: Canakinumab
Number analyzed (Participants) | 5 | 6 | 5 | 34
hours | 539 (47.1) | 578 (145) | 474 (93.6) | 736 (243)

23. Secondary Outcome: Apparent Clearance of Canakinumab From Plasma (CL/F)
Time Frame: Day 1, pre-dose and 1, 3, 6 and 8 hours post-dose (Part A only), Day 2, 4, 8, 15, 29, 57, 85 and 126.
Population: Pharmacokinetic analysis set, where data were available.
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | Part A: Canakinumab 150 mg | Part A: Canakinumab 300 mg | Part A: Canakinumab 600 mg | Part B: Canakinumab
Number analyzed (Participants) | 5 | 6 | 5 | 33
mL/hr | 9.58 (3.08) | 9.66 (2.03) | 13.3 (4.27) | 8.65 (3.02)

24. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase (Vz/F)
Time Frame: Day 1, pre-dose and 1, 3, 6 and 8 hours post-dose (Part A only), Day 2, 4, 8, 15, 29, 57, 85 and 126.
Population: Pharmacokinetic analysis set, where data were available.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Part A: Canakinumab 150 mg | Part A: Canakinumab 300 mg | Part A: Canakinumab 600 mg | Part B: Canakinumab
Number analyzed (Participants) | 5 | 6 | 5 | 33
mL | 7320 (1870) | 8060 (2830) | 8930 (3000) | 8910 (4070)

ADVERSE EVENTS:
Arm/Group | Part A: Canakinumab 150 mg | Part A: Canakinumab 300 mg | Part A: Canakinumab 600 mg | Part A: Placebo | Part B: Canakinumab | Part B: Placebo | Part B: Naproxen
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 1/6 | 1/5 | 0/45 | 4/47 | 4/53
Other Adverse Events (participants affected / at risk) | 4/6 | 4/7 | 3/6 | 3/5 | 17/45 | 25/47 | 26/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Canakinumab 150 mg (N=6) | Part A: Canakinumab 300 mg (N=7) | Part A: Canakinumab 600 mg (N=6) | Part A: Placebo (N=5) | Part B: Canakinumab (N=45) | Part B: Placebo (N=47) | Part B: Naproxen (N=53)
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Canakinumab 150 mg (N=6) | Part A: Canakinumab 300 mg (N=7) | Part A: Canakinumab 600 mg (N=6) | Part A: Placebo (N=5) | Part B: Canakinumab (N=45) | Part B: Placebo (N=47) | Part B: Naproxen (N=53)
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Retinal tear (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 3 | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 4 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 3
Cellulitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 4 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 2 | 7
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 1 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 3
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 4 | 6 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 4
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 2
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 5 | 6 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 3 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.